CLINICAL TRIAL: NCT06082219
Title: Ulcer Bleeding After Band Ligation of Esophageal Varices:Risk Factors and Prognosis
Brief Title: Ulcer Bleeding After Band Ligation of Esophageal Varices
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amna Esmail Mohamed Tamam, doctor, Assiut University
Other Study IDs: Post banding ulcer bleeding
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Esophageal Varices
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Primary Outcomes:

assessment of incidence , risk factors and prognosis of post-banding ulcer bleeding following EVL in patients with liver cirrhosis.

Secondary Outcomes:

minimize post-banding ulcer bleeding

DETAILED DESCRIPTION:
Esophageal variceal bleeding represents the most vital complication among patients with liver cirrhosis at rate of 5-15% per year. Endoscopic variceal ligation (EVL), either used as therapeutic in emergency or as prophylactic, is one of the best modalities used in EV treatment. The procedure is effective and generally safe. After banding, a superficial ulcer is formed, which usually heals in 2-3 weeks. The main complications of variceal banding are pain, dysphagia, fever, bleeding during the procedure and post banding ulcer bleeding (PBUB). The prevalence of PBUB is reported to be 3.6-15% . Rebleeding can be fatal, and is mainly resulted from early spontaneous slippage of the rubber bands, before occlusion of the varix with a mature thrombus, leaving an unhealed ulcer . The time frame of variceal rebleeding can be divided into very early rebleeding (within 5 days of acute bleeding), early rebleeding (within 6 weeks of acute bleeding), and delayed rebleeding. Previous reports showed that early rebleeding ranged from 30% to 40% within the first 6 weeks, and was significantly associated with the risk of death within 6 weeks. Therefore, the aim of this research is assessment of incidence , risk factors and prognosis of post-banding ulcer bleeding following EVL in patients with liver cirrhosis, in order to minimize post-banding ulcer bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age is 18 years or above.
2. Patient who are diagnosed with esophageal varices by upper endoscopy.
3. Patient who are fit for surgery to undergo endoscopic banding procedure.

Exclusion Criteria:

1. Pediatric patients.
2. patient refuse to participate at this study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients having esophageal varices who will undergo endoscopic banding will be included
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
assessment of incidence , risk factors and prognosis of post-banding ulcer bleeding following EVL in patients with liver cirrhosis. | Baseline
  assessment of incidence , risk factors and prognosis of post-banding ulcer bleeding following EVL in patients with liver cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Amna Esmail Mohamed Tammam, Principal Investigator — Assiut University; Essam Abdelmonem Sadek, Study Director — Assiut University; Muhammad Abbas Said El-Masry, Study Director — Assiut University